CLINICAL TRIAL: NCT01613391
Title: Effect of Roux-en-Y Gastric Bypass Versus Laparoscopic Adjustable Gastric Band Operations on Resistin, Apelin and Visfatin Peptides
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Muhammet Ferhat CELİK, Medical Doctor, Istanbul University
Other Study IDs: IU-BS-2012-RAV
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Morbid Obesity
Keywords: Visfatin; Resistin; Apelin; roux-en-y gastric bypass; laparoscopic adjustable gastric banding; morbid obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- RYGBP: Patients underwent Roux-en-Y Gastric Bypass for morbid obesity.
- LAGB: Patients underwent Laparoscopic Adjustable Gastric Banding for morbid obesity.

SUMMARY:
This study aimed to measure, compare apelin, resistin, visfatin levels in patients underwent to RYGBP, LAGB and their relation with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of morbid obesity
* Being underwent LAGB or RYGBP

Exclusion Criteria:

* Having prior abdominal surgery history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Morbidly obese 15 patients underwent LAGB and 15 patients underwent RYGBP
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)